CLINICAL TRIAL: NCT02646241
Title: Biopsy Protocol of Upper Gastrointestinal Subepithelial Tumors:Diagnostic Accuracy of EUS-FNB Versus Unroofing Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2015-1033
Record Dates: First submitted 2016-01-01; First posted 2016-01-05 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Upper Gastrointestinal Subepithelial Tumors
Keywords: stomach neoplasm; biopsy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unroofing biopsy (Experimental)
  Interventions: Procedure: unroofing biopsy
- EUS-FNB (Active Comparator)
  Interventions: Procedure: EUS-FNB(endoscopic ultrasonography guided fine needle biopsy)

INTERVENTIONS:
Procedure: unroofing biopsy — Unroofing biopsy menas that the mucosa is resected with endoscopic mucosal resection and biopsies are done repeatedly for the exposed tumor with a conventional forcep. It will be performed for the patients with a suspected upper gastrointestinal subepithelial tumor after EUS-FNB. After unroofing biopsy, the final histopathological result will be used to determine diagnostic accuracy.
  Arms: unroofing biopsy
Procedure: EUS-FNB(endoscopic ultrasonography guided fine needle biopsy) — EUS-FNB will be performed for the same patients who have a gastrointestinal subepithelail tumor before unroofing biopsy. EUS-FNB is called when the tissue is obtained by puncutre of a tumor, the tissue whithin the lumen of the fine needle being detached by rotatin, and the needle withdrawn. The pathological result will be also used to compare diagnostic accuracy between EUS-FNB & unroofing biopsy.
  Arms: EUS-FNB

SUMMARY:
To increase the diagnostic accuracy of subepithelial tumors, larger tissue samples are required. It is difficult to obtain adequate tissue samples. There were several biopsy methods to obtain tissue samples. Pathological examination would include mitosis counts, particularly in hypoechoic subepithelial tumors located in the 4th layer of the gastric wall, where differentiation between leiomyoma of benign nature and gastrointestinal stromal tumor (GIST) of malignant potential is essential.

So We hypothesize that unroofing biopsy is an more appropriate method than EUS-FNB(endoscopic ultrasonography guided fine needle biopsy). We will compare diagnostic accuracy and complications between EUS-FNB & unroofing biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 19 years old and younger than 80 years old
* Suspected upper gastrointestinal subepithelial tumors(≥15mm, ≤35mm) that were originated from muscularis propria layer on endoscopic ultrasonography(EUS)

Exclusion Criteria:

* Patient who had bleeding tendency
* Any previous surgery on esophagus, stomach or duodenum
* Patients who can not be underwent sedated endoscopy
* Gastrointestinal subepithelial tumor that was not origianted from muscularis propria layer on EUS
* Constrast related allergic disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy | within 7 days
  We will compare between diagnostic accuracy of EUS-FNB & unroofing biopsy using final histopathological result.

SECONDARY OUTCOMES:
number of complications of procedure | within 7 days
accuracy of malignant potential on contrast enhanced EUS | within 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Park JC, Jo JH, Kim EH, Shin SK, Lee SK, Lee YC. Prospective comparative study of endoscopic ultrasonography-guided fine-needle biopsy and unroofing biopsy. Dig Liver Dis. 2019 Jun;51(6):831-836. doi: 10.1016/j.dld.2019.01.028. Epub 2019 Feb 19. PMID 30872087